CLINICAL TRIAL: NCT03555175
Title: Value Eccentric and Proprioception Exercise Into the Injury Effect in Amateur Football
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Daniela Fernández, Physiotherapist, University of Alcala
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CEIM/HU/2018/06
Record Dates: First submitted 2018-05-05; First posted 2018-06-13 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Hamstring Injury
MeSH Terms: interventions — Proprioception; Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group one (Other): This participants group must do eccentric exercise for 12 weeks
  Interventions: Other: Eccentric exercise
- Group two (Other): This participants group must do proprioception exercise for 12 weeks
  Interventions: Other: Proprioception
- Group 3 (Other): This participants group mustn't do exercise extra
  Interventions: Other: Control group

INTERVENTIONS:
Other: Eccentric exercise — The group make hamstring eccentric exercise. The participants have to do 12 serie of 6 repeats
  Arms: Group one
Other: Proprioception — The group have to do three kinds of exercise in a inestable area during 15 second in 2 repeats for each one
  Arms: Group two
Other: Control group — Any exercise
  Arms: Group 3

SUMMARY:
This study evaluates the injury in amateur football, adding different excercise into the habitual practice. There are three groups, one of them do eccentric excercise, another group doing proprioception exercise and the last group don´t do any exercise.

DETAILED DESCRIPTION:
There are three group with 10 participants each one. The group one will do hamstring eccentric exercise 12 series per 6 repeats. The group two will do three proprioception exercise 2 series per exercise and leg. And third group won't have add some exercise to their normal training.

All participants will do the exercises during 12 weeks. Before this 12 weeks they will be valuation with different tests, and this tests will have to repeat after this 12 weeks and 3 weeks after finish the exercises.

ELIGIBILITY:
Inclusion Criteria:

* Training three times per week, add match day
* More than two years of experience
* Not be injured
* Not having been operated on the lower extremity

Exclusion Criteria:

-

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-06-15 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Y-Test (star test) | Three time. Before intervention, at the end and three weeks post-intervention
  Stability test. The participants have to do three directions in the test antrior, posteromedial and posterolateral. And they have to touch with their toe. And the investigator will measure the distance between his support foot and his moving foot
Vertical Jump test | Three times. Before intervention, at the end and three weeks post-intervention
  5 practice jumps with the hands in the hip, and we record this jumps. The investigator will measure distance between the participants feet and the floor in the upper point

SECONDARY OUTCOMES:
Weight | Before start
  Scales [kilogram]
Years | Before start
  Year of birth. Number
Height | Before start
  Metre
Years playing football | Before start
  Number of years. Number
Position in the team | Before start
  name of position player. Name

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Fernandez, Principal Investigator — The University of Alabama in Huntsville
Locations (1):
- Daniela Fernandez, Getafe, Madrid, Spain